CLINICAL TRIAL: NCT01386398
Title: Progression Free Survival (PFS) Comparison Between Suberoylanilide Hydroxamic Acid (SAHA, Vorinostat TM) in Combination With Bortezomib (Velcade TM) and SAHA Alone in Refractory or Recurrent Advanced CTCL. A Randomized Study.
Brief Title: Vorinostat With or Without Bortezomib in Treating Patients With Refractory or Recurrent Stage IIB, Stage III, or Stage IV Cutaneous T-Cell Lymphoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company withdrew interest
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-21082; EORTC-21082; EU-21116; EUDRACT-2009-011021-13
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Lymphoma
Keywords: stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — Bortezomib; Vorinostat

INTERVENTIONS:
Drug: bortezomib
Drug: vorinostat
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Vorinostat and bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether vorinostat is more effective when given alone or when given together with bortezomib in treating patients with refractory or recurrent cutaneous T-cell lymphoma.

PURPOSE: This randomized phase III trial is studying how well vorinostat works when given alone compared with vorinostat given together with bortezomib in treating patients with refractory or recurrent stage IIB, stage III, or stage IV cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if the combination of bortezomib plus vorinostat (SAHA) is more effective than vorinostat alone, in terms of prolonging progression-free survival, in patients with stage IIB-IV cutaneous T-cell lymphoma who have failed prior therapy.

Secondary

* To determine the overall survival of these patients.
* To determine the response rate in these patients.
* To determine the time to progression in these patients.
* To determine the duration of response in these patients.
* To determine the incidence of second cancers in these patients.
* To determine the acute and late toxicity of this regimen in these patients.
* To determine if translational research may provide insight into disease mechanism and identify biomarkers useful for prediction of treatment response. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to type of cutaneous T-cell lymphoma (mycosis fungoides vs erythrodermic mycosis fungoides/Sézary syndrome), number of prior chemotherapy regimens (1 vs ≥ 2), and country. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral vorinostat (SAHA) once daily in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive bortezomib IV on days 1, 4, 8, and 11 and oral vorinostat once daily on days 1-14. Treatment repeats every 21 days until progression or unacceptable toxicity.

Blood and tissue samples are collected periodically for translational research to provide insight into disease mechanism and identify biomarkers useful for prediction of treatment response.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months until disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced cutaneous T-cell lymphoma (CTCL), including its variants mycosis fungoides and Sézary syndrome

  * Stage IIB-IV disease
* Relapsed or refractory disease, including any of the following:

  * Patients with clinical progression following EORTC-21081 protocol treatment
  * Intolerant to ≥ 1 prior intravenous chemotherapy, including denileukin diftitox, antibodies or antibody conjugates, or any other systemic therapy
* No CNS involvement

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Absolute neutrophil count > 1.5 x 10^9/L*
* Platelet count > 100 x 10^9/L*
* Hemoglobin > 9 g/dL*
* WBC > 3 x 10^9/L*
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)*
* AST and ALT ≤ 3 times ULN (in case of liver infiltration ≤ 5 x ULN)*
* Serum creatinine ≤ 2.0 mg/dL*
* Calculated creatinine clearance ≥ 60 mL/min
* Electrolytes (including potassium and magnesium) ≤ 1 times ULN*
* Not pregnant or nursing prior to the first dose of study treatment and until 4 weeks after the last study treatment
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* Able to swallow capsules and is able to take or tolerate oral medication on a continuous basis
* No New York Heart Association class III-IV disease
* None of the following known conditions:

  * Infectious disease
  * Autoimmune disease
  * Immunodeficiency
* No known or active HIV and/or hepatitis A, B, or C infection
* No NCI CTC grade 1 peripheral sensory neuropathy with pain or peripheral sensory or motor neuropathy ≥ grade II
* No other malignancy within the past 5 years
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule NOTE: *Patients with a buffer range from the normal values of +/- 5% for hematology and +/- 10% for biochemistry are acceptable, except for renal function.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Must have completely recovered from previous treatment toxicity
* No prior splenectomy or splenic irradiation
* No prior bortezomib and/or histone deacetylase inhibitors (including vorinostat [SAHA])
* More than 4 weeks since prior chemotherapy, immunotherapy, radiotherapy, or surgery

  * In case of clear progression during previous treatment, 2 weeks of wash-out is enough
* No concurrent chemotherapy, immunotherapy, radiotherapy, or surgery (except biopsies)
* No concurrent steroid (prednisone or equivalent) dose > 20 mg/day

  * Prednisone ≤ 20 mg/day for treatment of disorders other than CTCL allowed
* No concomitant use of other histone deacetylase inhibitors (e.g., valproic acid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Response rate
Time to progression
Duration of response
Second cancers
Acute and late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Luis Ortiz-Romero — Hospital Universitario 12 de Octubre

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956